CLINICAL TRIAL: NCT00519688
Title: A Phase II Study of Tegafur/Uracil(UFUR) Plus Thalidomide for the Treatment of Advanced or Metastatic Hepatocellular Carcinoma (HCC)
Brief Title: UFUR Plus Thalidomide for Advanced Hepatocellular Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 940813; TTY-TU0510
Record Dates: First submitted 2007-08-22; First posted 2007-08-23 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Hepatocellular Carcinoma
Keywords: tegafur; thalidomide; advanced hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Thalidomide; Tegafur

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Thalidomide plus Tegafur/Uracil1 (Experimental): Thalidomide plus Tegafur/Uracil
  Interventions: Drug: Thalidomide; Drug: Tegafur/Uracil

INTERVENTIONS:
Drug: Thalidomide — 100 mg, BID
  Other Names: Thado
Drug: Tegafur/Uracil — 125 mg/m2, based on tegafur, BID
  Other Names: UFUR

SUMMARY:
We hypothesize that combination of tegafur/uracil(UFUR) and thalidomide, both of which have been shown to be active in some HCC patients,may be a highly useful regimen for the treatment of advanced HCC. There are several rationales underlying this combination. First, anti-angiogenesis therapy may improve the efficacy of chemotherapy by normalizing the abnormal vasculature in tumors, and thus improving the delivery of chemotherapeutic agents to the tumor cells. Second, chemotherapeutic drugs given in a low-dose, un interrupted, and protracted way can induce anti-tumor effect through the anti-angiogenesis activity (so-called"metronomic chemotherapy"). The efficacy of metronomic chemotherapy can be suppressed by VEGF/VEGFR signaling pathways and thus can bo further potentiated by agents blocking those survival signals of endothelial cell. In this regard, tegafur/uracil appears to be a good candidate for metronomic chemotherapy because tegafur/uracil and its metabolites bave already been shown to inhibit angiogenesis in several pre-clinical models.

DETAILED DESCRIPTION:
Thalidomide, a glutamic acid derivative first developed in 1950s, was marketed as a sedative, tranquilizer, and antiemetic for morning sickness. It was withdrawn from the European and Canadian markets in early 1960s because of its teratogenic effects. In recent years, thalidomide is emerging as a novel treatment for cancer because of its anti-angiogenic properties. The clinical efficacy has been demonstrated in various types of human cancers, including HCC.

Tegafur and uracil is a composite drug, which has been marketed as UFT® in Japan and marketed as UFUR® in Taiwan. Tegafur, a prodrug of 5-FU, is easily absorbed though the gastrointestinal tract slowly metabolized to 5-FU mainly in liver. Uracil is an inhibitor of dihydropyrimidine dehydrogenase (DPD), the rate-limiting enzyme of 5-FU degradation. Therefore, tegafur/uracil is expected to maintain a stably high concentration in liver and in circulation. Tegafur/uracil has been approved for the indications of advanced gastric cancer and colorectal cancer. In several phase II studies conducted in Japan, tegafur/uracil induced a response rate of 0 to 17% in advanced HCC patients.

We hypothesize that combination of tegafur/uracil and thalidomide, both of which have been shown to be active in some HCC patients, may be a highly useful regimen for the treatment of advanced HCC. There are several rationales underlying this combination. First, anti-angiogenesis therapy may improve the efficacy of chemotherapy by normalizing the abnormal vasculature in tumors, and thus improving the delivery of chemotherapeutic agents to the tumor cells. Second, chemotherapeutic drugs given in a low-dose, un-interrupted, and protracted way can induce anti-neoplasm effect through the anti-angiogenesis activity. What so-called "metronomic chemotherapy" is based on direct targeting of the activation, growth, and proliferation of vascular endothelial cells by cytotoxic chemotherapeutic agents. The anti-angiogenesis effect of metronomic chemotherapy is suppressed by VEGF/VEGFR signaling pathways and thus can be further potentiated by agents blocking those survival signals of endothelial cells. In this regard, tegafur/uracil appears to be a good candidate for metronomic chemotherapy because tegafur/uracil and its metabolites have already been shown to inhibit angiogenesis in several pre-clinical models.

The combination of tegafur/uracil and thalidomide has clinical advantages for patients with HCC. Both drugs are orally active, thus are convenient to be given on an out-patient basis. More importantly, the low and non-overlapping toxicity profiles of the two drugs make the combination relatively safe in patients of HCC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed HCC or HBC/HCV carrier with hepatic tumor of α-FP>400 Stage IV dis. By AJCC KPS>70% Age>18 Liver function reserves:Child-Pugh Class A, ALT<5xUNL, Bil-T<1.5xUNL WBC>4000 or ANC>1500, PLT>75K, Cr<1.5xUNL Previous local therapy completed 6wks

Exclusion Criteria:

* Concurrent corticosteroids Previous exposure to C/T, Thalidomide CNS metastasis Concomitant illness: active infection, >NCIG2 neuropathy, Hx of seizures Organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2006-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the overall response rate of UFUR and thalidomide in the treatment of advanced HCC by RECIST criteria | Confirmed response within 4 weeks

SECONDARY OUTCOMES:
To determine the disease stabilization rate. | 2 to 3 months
To assess the progression- free survival and overall survival. | 2 to 3 years
To establish the safety profile. | Additional 4 months after stopping the investigational drugs
  Toxicity criteria based on CTC-AE version 3

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Hung Hsu, M.D. Ph.D., Study Chair — Department of Oncology, National Taiwan University hospital
Locations (1):
- Department of Oncology , National Taiwan University Hospital, Taipei, Taiwan